CLINICAL TRIAL: NCT00429182
Title: Phase II Study of Purging of Circulating Tumor Cells (CTCs) From Metastatic Breast Cancer Patients
Brief Title: Purged Circulating Tumor Cells (CTCs) From Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0280
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer; Metastatic Breast Carcinoma; Invasive Breast Carcinoma
Keywords: Breast Cancer; breast carcinoma; Carboplatin; Paraplatin; Cyclophosphamide; Neosar; Cytoxan; Thiotepa; Purged Autologous Stem Cells; Circulating Tumor Cells; CTCs
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Carboplatin; Cyclophosphamide; Thiotepa; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High-dose chemotherapy (Experimental): Carboplatin + Cyclophosphamide + Thiotepa
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Thiotepa; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Carboplatin — Target Area Under the Curve (AUC) of 20, then divided into 4 doses given by vein (IV) days -6, -5, -4, -3 prior to stem cell infusion.
  Other Names: Paraplatin
Drug: Cyclophosphamide — 1.5 gm/m^2 by vein days -6, -5, -4, -3 prior to stem cell infusion.
  Other Names: Cytoxan; Neosar
Drug: Thiotepa — 120 mg/m^2 by vein days -6, -5, -4, -3 prior to stem cell infusion.
Procedure: Stem Cell Transplant — Stem Cell Transplant on Day 0.
  Other Names: SCT; Autologous hematopoietic stem cell transplantation; AHST

SUMMARY:
The goal of this clinical research study is to learn the relationship of high-dose chemotherapy (HDCT) and circulating tumor cells (CTCs) in controlling metastatic breast cancer. The study also will investigate the role of CTCs in breast cancer.

DETAILED DESCRIPTION:
Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die. Carboplatin and thiotepa are designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die. Mesna is designed to prevent toxicities from cyclophosphamide. Granulocyte colony-stimulating factor (G-CSF or GCSF) is designed to help your white blood count recover after transplant.

If you are found to be eligible to take part in this study, you will be given G-CSF twice a day through a needle under the skin (subcutaneous injection), on Days 1-5. On Day 5, stem cell collection will begin. You will have a catheter placed into a vein in your chest. A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your physician will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

If further shrinkage of tumor is needed, the doctor may use chemotherapy combined with G-CSF described above. Your doctor will explain this procedure to you in more detail, and you will be asked to sign a separate consent form for this procedure.

Blood will be removed from your body through the catheter and passed through a machine that separates the stem cells from the other cells. The stem cells will be frozen for storage, and the blood will be returned to your body. This 3-hour process is called apheresis. The process will be done once a day for 1-6 days until enough stem cells are collected. Blood ( about 4 teaspoons) will be collected at the first Apheresis to have as a comparison sample to check for any breast cancer leftover in the blood.

The collected blood cells will go through a filter to select out the blood stem cells and the CTCs will be left behind.

Blood (about 2 tablespoons) will be drawn daily during peripheral blood stem cell collection.

On Days 6, 5, 4, and 3 before the transplant, you will receive cyclophosphamide, mesna, thiotepa, and carboplatin through a needle in your vein. Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 0, your stem cells will be transplanted. Stem cells will go through a device to remove the breast cancer cells. If the bone marrow is collected because there was not enough stem cells, researchers will not treat the bone marrow to remove breast cancer cells. Collected breast cancer cells will be studied to understand the biological role of these cancer cells.

After the transplant, G-CSF will be given through a needle under your skin until the white blood cell count is normal for 3 days in a row.

Blood (about 2 tablespoons) will be drawn daily after the transplant while you are still in the hospital. You are expected to remain in the hospital for 3 weeks. Once you are released from the hospital, you will have blood (about 2 tablespoons) drawn for routine tests every week until your cell counts recover.

Five (5) weeks after your transplant, if your doctor thinks it is needed, you will have radiation therapy, hormonal therapy, or receive trastuzumab.

At Months 1, 3, 6, 9, 12, 16, 20, and 24 after the transplant, your complete medical history will be recorded, and you will have a physical exam. You will have a chest X-ray and bone scan. If your doctor thinks it is needed, you will have an x-ray of hot spots which are areas that show positive on the bone scan. If your doctor thinks it is needed, you may have a CT scan of the head, a mammogram, or a breast ultrasound performed. At Months 1 and 3 after the transplant, you will have a PET/CT scan. At Months 6, 9, 12, 16, 20, and 24 after the transplant, you will have a CT scan of the chest and abdomen then as needed to check the status of the disease. Blood (about 2 teaspoons) will be drawn to measure cancer markers and CTCs.

While on study you must notify the doctor of any new drugs you are taking.

This is an investigational study. The transplant is not FDA approved. The drugs G-CSF, cyclophosphamide, carboplatin, and thiotepa are all approved by the FDA and commercially available. The CliniMACS device is not commercially available or FDA approved. The CliniMACS device is being used in research only and will be provided free of charge. Up to 70 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 55 years old
2. Metastatic breast carcinoma.
3. Histological confirmation of invasive breast carcinoma
4. Complete or partial response to pre-transplant standard-dose chemotherapy, or hormonal therapy. For bone disease, stable disease (SD) is allowed.
5. Patient must have tumor assessed for estrogen-receptor (ER) and progesterone-receptor (PR).
6. Persistent detectable or non-detectable CTCs by Veridex Technology after completion of standard therapy.
7. Zubrod performance status 0 or 1.
8. Patients must have adequate hematological parameters (White Blood Count/WBC >= 3,000/mm3; platelet count >= 100,000/mm3)
9. Adequate renal function (serum creatinine <= 1.5mg/dl)
10. Adequate liver function (total bilirubin, serum glutamate pyruvate transaminase (SGPT) <= 2 times normal).
11. Adequate cardiac function (Left ventricular ejection fraction (LVEF)>= 50%).
12. Adequate pulmonary function (Carbon Monoxide Diffusing Capacity (DLCO)>= 50% of predicted value).
13. Females of childbearing (women who are post-menopausal < 1 year, not surgically sterilized, or not abstinent) potential must use adequate contraception.
14. Patients must sign an informed consent.

Exclusion Criteria:

1. Prior HDCT with Autologous hematopoietic stem cell transplantation (AHST) in adjuvant setting.
2. History or presence of brain/leptomeningeal metastasis.
3. History of other malignancies except cured non-melanoma skin cancer or cured cervical carcinoma in situ.
4. Presence of other severe medical illnesses or conditions. Severe heart disease, (myocardial ischemia, myocardial infarction, etc.) Pulmonary disease (COPD, asthma,etc). Renal failure and hepatic failure.
5. Clinically significant active infections (patient requiring IV antibiotics, uncontrolled infections, or hospitalized due to infections).
6. HIV infection.
7. Pregnant or lactating women.
8. Medical, social or psychologic factors which would prevent the patient from receiving or cooperating with the full course of therapy or understanding the informed consent procedure.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 27, 2007 to July 25, 2011. All Recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- High-dose Chemotherapy: Carboplatin + Cyclophosphamide + Thiotepa
  Carboplatin : Target area under the curve (AUC) of 20, then divided into 4 doses given by vein (IV) days -6, -5, -4, -3 prior to stem cell infusion.
  Thiotepa : 120 mg/m^2 by vein days -6, -5, -4, -3 prior to stem cell infusion.
  Stem Cell Transplant : Stem Cell Transplant on Day 0.
  Cyclophosphamide : 1.5 gm/m^2 by vein days -6, -5, -4, -3 prior to stem cell infusion.
Period: Overall Study
Arm/Group | High-dose Chemotherapy
Started | 32
Completed | 25
Not Completed | 7
Not completed — Not evaluable, Disease Progression | 2
Not completed — Not eligible | 5

BASELINE CHARACTERISTICS:
Groups:
- High-dose Chemotherapy: Carboplatin + Cyclophosphamide + Thiotepa
  Carboplatin : Target AUC of 20, then divided into 4 doses given by vein (IV) days -6, -5, -4, -3 prior to stem cell infusion.
  Thiotepa : 120 mg/m^2 by vein days -6, -5, -4, -3 prior to stem cell infusion.
  Stem Cell Transplant : Stem Cell Transplant on Day 0.
  Cyclophosphamide : 1.5 gm/m^2 by vein days -6, -5, -4, -3 prior to stem cell infusion.
Arm/Group | High-dose Chemotherapy
Number analyzed (Participants) | 32
Age Continuous [Median (Full Range); unit: years] | 44 [29 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction in CTCs Following High-dose Chemotherapy With Purged Autologous Stem Cell Products
Description: Number of circulating tumor cells (CTCs) measured at one month post autologous hematopoietic stem cell transplantation (AHST), considered both as longitudinal values and compared to the baseline number of CTCs.
Time Frame: Baseline to 1 month post AHST
Population: Twenty-one participants provided blood samples for the enumeration of CTCs, before apheresis (baseline) and at one month after AHST.
Measure: Number; unit: participants
Arm/Group | High-dose Chemotherapy
Number analyzed (Participants) | 21
participants | 9

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Kaplan-Meier estimate of the median time from randomization to death from any cause or first observed disease progression. PFS time measured in months.
Time Frame: Overall study (baseline to disease progression)
Population: Six participants were not evaluable for outcome assessment.
Measure: Median (Full Range); unit: months
Arm/Group | High-dose Chemotherapy
Number analyzed (Participants) | 26
months | 10.6 [1 to 16.4]

ADVERSE EVENTS:
Time Frame: 4 years and 5 months
Arm/Group | High-dose Chemotherapy
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Chemotherapy (N=32)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Chemotherapy (N=32)
Nausea (Gastrointestinal disorders) | 27
Diarrhea (Gastrointestinal disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No